CLINICAL TRIAL: NCT04226001
Title: Impact of a Carrier (Infection, Colonization) of Highly Bacteria Resistance on the Patient's
Brief Title: Impact of a Carrier (Infection, Colonization) of Highly Bacteria Resistance on the Patient's Quality of Life Hospital Environment
Acronym: QALYBHRe
Status: Withdrawn | Type: Observational
Why Stopped: Coordinator departure
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0022; 2019-A00074-53 (Other: ID-RCB)
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients screened for carriers infected or colonized by emerging highly resistant bacteria.
  Interventions: Other: Quality of life questionnaire

INTERVENTIONS:
Other: Quality of life questionnaire — Quality of life questionnaire

SUMMARY:
The quality of life of carriers detected infected or colonized by emerging highly resistant bacteria (BHRe) following the implementation of specific hygiene measures during the discovery of the microorganism has been little studied. To date, there have been no studies to determine the quality of life (QoL) in France of patients with hospitalized HBHRD.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old
* Have a positive BHRe screening during the hospital stay and / or have a positive BHRe clinical sample during the hospital stay
* Conscious patients
* All types of stays in the hospital sector
* All pathologies

Exclusion Criteria:

* Known patients with BHRe before hospitalization
* PCH immediately upon admission (history of hospitalization abroad, patients contacted during a previous hospitalization)
* Cognitive problem
* Patients not proficient in French (requiring an interpreter)
* Patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients infected or colonized by emerging highly resistant bacteria.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Impact of the implementation of Complementary Hygiene Precautions following a carrier of emerging highly resistant bacteria on the quality of life of hospitalized patients | 12 months
  Measurement of the decrease in utility corresponding to the deterioration of the QOL of patients since the implementation of the Additional Hygiene Precautions (PCH) following the discovery of their emerging highly resistant bacteria (BHRe).

CONTACTS AND LOCATIONS:
Overall Officials: David NARBEY, MD, Principal Investigator — Hospices Civils de Lyon